CLINICAL TRIAL: NCT02951663
Title: Evaluation of Body Composition and Metabolism Following Bariatric Surgery, Effects of a Protein Supplement: A Feasibility Study
Brief Title: Protein Supplementation Post Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-0529
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein Supplement (Experimental): Ready to drink blinded protein supplement
  Interventions: Dietary Supplement: Protein
- Control (No Intervention): Control group

INTERVENTIONS:
Dietary Supplement: Protein
  Arms: Protein Supplement

SUMMARY:
Purpose: To evaluate adherence, tolerability, and total protein intake in bariatric surgery patients provided with ready-to-drink protein supplements, and to evaluate the effects of supplementation on body composition, metabolism, and health outcomes.

Participants: Patients scheduled to under go bariatric surgery aged 18-70 years old. Participants will be included if they agree to comply with the study protocol, are free of medical conditions that may contraindicate participation, and do not plan to become pregnant during the study.

Procedures (methods): Participants will complete five laboratory visits for the current study (pre-screening (visit 1), baseline testing (visit 2), and return visits at 3 weeks (visit 3), 12 weeks (visit 4), and 24 weeks (visit 5) post-surgery). The treatment group will be given a 12 week supply of a high protein, low-carbohydrate, low-fat supplement to be taken once daily during days 3-7 post-surgery, and twice daily weeks 2-12. The treatment group will follow standard of care recommendations put forth by the physician-nutritionist team, but using the provided protein supplement to meet recommendations. The control group will be asked to follow the standard of care recommendations from the physician-nutritionist team.

The primary study endpoints will be adherence, tolerability, and total protein intake in bariatric surgery patients provided with a 12-week supply of ready-to-drink protein supplements. Secondary outcomes will evaluate the effect of a protein supplement on body composition (lean mass, fat mass, percent body fat, visceral fat, muscle thickness), resting metabolic rate, clinical and endocrine blood values, functional fitness, and responses to questionnaires evaluating mood, satiety, functional independence, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled for weight loss surgery
* Participant agrees to abstain from extraneous supplementation with creatine, β-hydroxy β-methylbutyrate, carnosine, beta-alanine, taurine, or any other supplement or prescription drug that may significantly influence body composition or metabolic rate
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing and able to comply with the protocol
* Participant agrees to abstain from using caffeine, tobacco, and alcohol for at least 24 hours before testing days
* Participant agrees to abstain from exercise 24 hours prior to each testing visit
* Participant is not currently pregnant and does not desire to become pregnant in the next six months

Exclusion Criteria:

* Physicians on the research team believe that a pre-existing condition may influence participant safety or study outcomes, including previously diagnosed cardiovascular, metabolic, renal, hepatic, or musculoskeletal disorders
* Participant is using, or has used one of the following dietary supplements within 8 weeks prior to enrollment: creatine, β-hydroxy β-methylbutyrate, carnosine, beta-alanine, taurine, or any other supplement or prescription drug that may significantly influence body composition or metabolic rate
* Participant is in, or has participated in another clinical trial within 4 weeks prior to enrollment
* Participant is pregnant or plans on becoming pregnant
* Participant has a known allergy or sensitivity to any ingredient in the test product (determined from health history questionnaire)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting gastrointestinal effects during use of supplementation | 12 weeks
  Tracked using a custom survey
Number of shakes consumed out of the total number of shakes provided | 12 weeks

SECONDARY OUTCOMES:
Body fat | 12 weeks
  measured using ultrasound
Lean body mass | 12 weeks
  measured using ultrasound
Metabolism (resting metabolic rate) | 12 weeks
Functional fitness (sit to stand test) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Exercise & Sport Science and GI Surgery UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch KR, Blue MNM, Trexler ET, Ahuja S, Smith-Ryan AE. Provision of ready-to-drink protein following bariatric surgery: An evaluation of tolerability, body composition, and metabolic rate. Clin Nutr. 2021 Apr;40(4):2319-2327. doi: 10.1016/j.clnu.2020.10.022. Epub 2020 Oct 23. PMID 33158590